CLINICAL TRIAL: NCT00372606
Title: An Evaluation of a Culturally- and Linguistically-Appropriate eHealth Portal to Facilitate Improved Diets, Increased Fitness-Levels, and Weight-Loss Among U.S. Hispanics
Brief Title: An Evaluation of a Culturally- and Linguistically-Appropriate Online Diet Program for U.S Hispanics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Responsible Party: Dirk Schroeder, DrTango
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 51759
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Hispanics; Online; Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

INTERVENTIONS:
Behavioral: Online MiDieta Diet and Weight Management Program for Hispanics

SUMMARY:
The purpose of this study is to conduct a randomized trial to rigorously test the efficacy of the MiDieta eHealth portal for weight loss among overweight, though otherwise healthy, members of the Hispanic community, many of whom may be members of collaborating managed care organizations.

DETAILED DESCRIPTION:
Obesity is a major and growing problem among U.S. Hispanics with serious implications for diabetes and other chronic disease risks. Current trends among youth suggest that disparities in obesity between minorities and non-Hispanic whites will amplify. Reducing such health disparities is a priority for federal, state and local governmental bodies and communities. Attaining these objectives will require interventions that are culturally- and linguistically appropriate. U.S. healthcare providers, however, have few culturally-appropriate tools and inadequate numbers of bilingual, trained healthcare professionals to address these challenges.

A culturally-appropriate weight-management portal, supported by bilingual Latina dietitians available for remote email counseling, offers an attractive mechanism for efficiently serving the underserved. MiDieta/MyDiet is the leading online diet, fitness and weight management portal for U.S. Hispanic/Latinos. MiDieta is bilingual (Spanish/English), based on Latino foods & habits and already available through dozens of media, hospital, and health plan websites. Thousands of Hispanics access MiDieta each week. Tommy Thompson recently selected MiDieta as one of the "20 most innovative health promotion and disease prevention applications" in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Women and men of Hispanic/Latino origin born in Mexico, Central or South America, the Caribbean, Spain or the United States
* Between 18 and 75 years of age
* BMI >/= 24.85
* Otherwise "healthy" individuals (lack of major medical/psychiatric/ or chronic problems/disease - with the exception of Type 2 diabetes and controlled hypertension)
* Not participating in other weight loss treatment programs and not planning on it for at least 12-16 more months
* Internet access at least once per week
* The participant has the ability to engage in at least light activity (walking, etc)

Exclusion Criteria:

* The participant has a continuous history of major medical or psychiatric problems (requiring continuous medication and/or close physician supervision)
* Diagnosis with Type 1 diabetes
* The participant is pregnant or planning a pregnancy within the next 16 months
* The participant is unable to participate in any exercise regimen
* The participant is currently participating in MiDieta
* The participant is currently participating in other weight loss programs or plans to in the next 12-16 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Weight loss

SECONDARY OUTCOMES:
Dietary behaviors
Fitness activities
Program acceptability by users

CONTACTS AND LOCATIONS:
Overall Officials: Dirk G Schroeder, ScD, MPH, Principal Investigator — DrTango, Inc.; Jessica L Malmad, MPH, Study Director — DrTango, Inc.
Locations (1):
- DrTango, Inc., Roswell, Georgia, United States